CLINICAL TRIAL: NCT01937559
Title: Topical Application of Tranexamic Acid in Joint Arthroplasty
Brief Title: Topical Tranexamic Acid (TXA) in Joint Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Hawkins Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00021253
Record Dates: First submitted 2013-08-30; First posted 2013-09-09 (Estimated); Results first posted 2020-05-05 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-04

CONDITIONS: Osteoarthritis; Hip Arthropathy; Shoulder Arthropathy
Keywords: tranexamic acid (TXA)
MeSH Terms: conditions — Osteoarthritis | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Topical Tranexamic acid (TXA) (Experimental): Tranexamic acid (TXA) applied topically
  Interventions: Biological: Tranexamic acid (TXA)
- Saline (Placebo Comparator): Normal saline
  Interventions: Drug: Normal saline
- Tranexamic acid (TXA) (Active Comparator): Tranexamic acid (TXA) administered intravenously
  Interventions: Biological: Tranexamic acid (TXA)

INTERVENTIONS:
Biological: Tranexamic acid (TXA) — 1.5g of TXA in 100ml normal saline solution
  Other Names: Cyklokapron
  Arms: Topical Tranexamic acid (TXA); Tranexamic acid (TXA)
Drug: Normal saline
  Arms: Saline

SUMMARY:
The objective of this study is to evaluate the efficacy of topical tranexamic acid (TXA) in decreasing blood loss following both shoulder arthroplasty and primary total hip arthroplasty. TXA functions to decrease blood loss by affecting the blood clotting system within the body. The investigators hypothesize that topical application of TXA prior to closure reduces postoperative bleeding as measured by absolute changes in postoperative hemoglobin levels and surgical drain output. In addition, use of topically applied tranexamic acid may reduce the need for transfusions, the rates of hematomas, infections, and length of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Shoulders: All adult patients over the age of 18 scheduled for a primary total arthroplasty or a primary reverse shoulder arthroplasty will be eligible for inclusion in the study.

Hips: All adult patients over the age of 18 scheduled for a primary total hip arthroplasty will be eligible for inclusion in the study.

Exclusion Criteria:

* allergy to TXA, refusal of blood products, preoperative use of anticoagulant therapy within 5 days of surgery, history of seizures, renal failure (creatine clearance <30ml/min), bleeding disorders, venous thromboembolism (deep vein thrombosis and/or pulmonary embolism), significant cardiac history (myocardial infarction, angina, stroke, lower limb ischemia), or perioperative anemia (hemoglobin <11g/dl in females and < 12g/dl in males).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Burnikel, MD, Principal Investigator — Steadman Hawkins Clinic of the Carolinas - Greenville Health System
Locations (1):
- Steadman Hawkins Clinic of the Carolinas - Greenville Health System, Greenville, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 122 patients were enrolled and randomized into one of two groups: tranexamic acid administered topically and saline administered topically (control). 61 patients were enrolled in each of the two groups. In addition, 66 patients who received tranexamic acid intravenously were retrospectively analyzed as a comparative group.
Groups:
- Topical Tranexamic Acid (TXA): Tranexamic acid (TXA): 1.5g of TXA in 100ml normal saline solution administered topically
- Saline (Control): Normal saline administered topically (control)
- Intravenous Tranexamic Acid (TXA): Current standard of care is Tranexamic acid (TXA) administered intravenously. This arm was added as a retrospective comparative group, thus these patients were not randomized during the original study.
Period: Overall Study
Arm/Group | Topical Tranexamic Acid (TXA) | Saline (Control) | Intravenous Tranexamic Acid (TXA)
Started | 61 | 61 | 66
Completed | 50 | 50 | 66
Not Completed | 11 | 11 | 0
Not completed — Physician Decision | 3 | 3 | 0
Not completed — Withdrawal by Subject | 6 | 4 | 0
Not completed — screen fail | 2 | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Topical Tranexamic Acid (TXA): TXA administered topically
  Tranexamic acid (TXA): 1.5g of TXA in 100ml normal saline solution administered topically
- Saline: Normal saline administered topically
- Total: Total of all reporting groups
Arm/Group | Topical Tranexamic Acid (TXA) | Saline | Intravenous Tranexamic Acid (TXA) | Total
Number analyzed (Participants) | 61 | 61 | 66 | 188
Age, Continuous [Mean (Full Range); unit: years] — Population: Several patients withdrew prior to primary endpoint being collected and thus were not included in analysis.
  years
    number analyzed (Participants) | 50 | 50 | 66 | 166
    (all) | 62 [35 to 86] | 65 [40 to 87] | 65 [35 to 83] | 64.2 [35 to 87]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Several patients withdrew prior to primary endpoint being collected and thus were not included in analysis.
  Participants
    number analyzed (Participants) | 50 | 50 | 66 | 166
    Female | 29 | 23 | 31 | 83
    Male | 21 | 27 | 35 | 83
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Several patients withdrew prior to primary endpoint being collected and thus were not included in analysis.
  Participants
    number analyzed (Participants) | 50 | 50 | 66 | 166
    Hispanic or Latino | 1 | 0 | 0 | 1
    Not Hispanic or Latino | 49 | 50 | 66 | 165
    Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Several patients withdrew prior to primary endpoint being collected and thus were not included in analysis.
  Participants
    number analyzed (Participants) | 50 | 50 | 66 | 166
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 5 | 4 | 5 | 14
    White | 45 | 46 | 61 | 152
    More than one race | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — Population: 22 patients were withdrawn prior to surgery (11 in the Topical tranexamic acid group and 11 in the saline group). These patients were not included in the analysis population due to their pre-operative withdrawal from the study.
  Participants
    United States: number analyzed (Participants) | 50 | 50 | 66 | 166
    United States | 50 | 50 | 66 | 166

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Blood Loss
Description: Blood loss will be calculated as the difference between the preoperative hemoglobin and the lowest postoperative hemoglobin during the hospital stay or the lowest postoperative hemoglobin prior to blood transfusion.
Time Frame: Duration of hospital stay, up to 4 days
Measure: Mean (Standard Deviation); unit: mL
Groups:
- Topical Tranexamic Acid (TXA): Tranexamic acid (TXA) administered topically
  Tranexamic acid (TXA): 1.5g of TXA in 100ml normal saline solution
- Intravenous Tranexamic Acid (TXA): Tranexamic acid (TXA) administered intravenously
Arm/Group | Topical Tranexamic Acid (TXA) | Saline | Intravenous Tranexamic Acid (TXA)
Number analyzed (Participants) | 50 | 50 | 66
mL | 1,062.88 (338.78) | 1,204.60 (403.61) | 933.92 (351.17)

2. Secondary Outcome: Number of Participants With Perioperative Blood Transfusions
Time Frame: Duration of hospital stay, up to 4 days
Measure: Number; unit: participants
Groups:
- Intravenous Tranexamic Acid (TXA): TXA administered intravenously
Arm/Group | Topical Tranexamic Acid (TXA) | Saline | Intravenous Tranexamic Acid (TXA)
Number analyzed (Participants) | 50 | 50 | 66
participants | 0 | 0 | 0

3. Secondary Outcome: Number of Blood Units Transfused
Time Frame: Duration of hospital stay, up to 4 days
Measure: Number; unit: blood units
Groups:
- Topical Tranexamic Acid (TXA): Topical Tranexamic acid (TXA)
  Tranexamic acid (TXA): 1.5g of TXA in 100ml normal saline solution
- Intravenous Tranexamic Acid (TXA): Intravenous Tranexamic acid (TXA)
Arm/Group | Topical Tranexamic Acid (TXA) | Saline | Intravenous Tranexamic Acid (TXA)
Number analyzed (Participants) | 50 | 50 | 66
blood units | 0 | 0 | 0

4. Secondary Outcome: Rate of Surgical Infections
Time Frame: Duration of hospital stay, up to 4 days
Measure: Count of Participants; unit: Participants
Groups:
- Topical Tranexamic Acid (TXA): Tranexamic acid (TXA)
  Tranexamic acid (TXA): 1.5g of TXA in 100ml normal saline solution
Arm/Group | Topical Tranexamic Acid (TXA) | Saline | Intravenous Tranexamic Acid (TXA)
Number analyzed (Participants) | 50 | 50 | 66
Participants | 0 | 0 | 0

5. Secondary Outcome: Length of Hospital Stay
Time Frame: Duration of hospital stay
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Topical Tranexamic Acid (TXA) | Saline | Intravenous Tranexamic Acid (TXA)
Number analyzed (Participants) | 50 | 50 | 66
days | 1.52 (0.61) | 1.64 (0.72) | 1.39 (0.63)

6. Secondary Outcome: Patient-reported Outcomes Scores, Including Euroqol-5D (EQ-5D), Global Rating of Change Scale (GRoC), and Single Alpha Numeric Evaluation (SANE).
Description: * Single Assessment Numeric Evaluation (SANE): A single question that asks "How would you rate your hip today as a percentage of normal (0% to 100% scale with 100% being normal)?" 0 indicates an abnormal shoulder, whereas 100% indicates a perfectly normal shoulder.
  * Euroqol-5D (EQ-5D): The EQ-5D is a patient-reported overall health questionnaire, with 100 indicating "The best health you can imagine" and 0 indicating "The worst health you can imagine."
  * Global Rating of Change Scale (GRoC): Provide a means of measuring self-perceived change in health status. The main purpose is to quantify the extent to which a patient has improved or deteriorated over time. The outcome is measured on a scale of -7 to 7, with -7 being the hip is "a very great deal worse from before surgery" and 7 being the hip is "a very great deal better from before surgery."
Time Frame: 6 months post-surgery
Population: Patient-reported outcomes were only collected for the two randomized patient groups (Topical tranexamic acid and saline). Patient-reported outcomes were not collected on the intravenous tranexamic acid group, as this group was added for retrospective comparison.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Topical Tranexamic Acid (TXA) | Saline
Number analyzed (Participants) | 50 | 50
score on a scale
  EQ-5D | 84.87 (13.69) | 80.15 (16.58)
  GRoC | 6.24 (0.91) | 5.54 (2.03)
  SANE | 89.06 (8.51) | 81.08 (21.61)

7. Secondary Outcome: Patient-reported Outcome Scores Including the Harris Hip Score and Western Ontario and McMaster Universities Arthritis Index (WOMAC)
Description: Harris Hip Score: Consists of 10 question items evaluating pain, function, absence of deformity, and range of motion. Scores range from 0-100 with higher scores representing less dysfunction and better outcomes, whereas lower scores represent more dysfunction and worse outcomes.
  Western Ontario and McMaster Universities Arthritis Index (WOMAC): Consists of 24 questions evaluating hip pain, stiffness and function. The score is normalized to a 100 point scale, where 0 indicates a poor outcome and 100 indicates the best outcome.
Time Frame: 6 months after surgery
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Topical Tranexamic Acid (TXA) | Saline
Number analyzed (Participants) | 50 | 50
score on a scale
  Harris Hip Score | 85.03 (15.90) | 79.95 (18.5)
  WOMAC | 14.64 (15.42) | 13.46 (11.23)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from date of surgery to 6 month follow-up. All adverse events from the date of surgery to the final 6 month follow-up were assessed and collected for each patient.
Arm/Group | Topical Tranexamic Acid (TXA) | Saline | Intravenous Tranexamic Acid (TXA)
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50 | 0/66
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50 | 0/66
Other Adverse Events (participants affected / at risk) | 4/50 | 0/50 | 4/66
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Topical Tranexamic Acid (TXA) (N=50) | Saline (N=50) | Intravenous Tranexamic Acid (TXA) (N=66)
ischemic stroke (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) — ischemic stroke reported 8 months after surgery
hematoma (Vascular disorders) | 2 (2) | 0 (0) | 1 (1)
deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 2 (2)
Aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-08): https://cdn.clinicaltrials.gov/large-docs/59/NCT01937559/Prot_SAP_000.pdf